CLINICAL TRIAL: NCT02431611
Title: Biomarker Feedback to Motivate Tobacco Cessation in Pregnant Alaska Native Women (MAW) - Phase 3 Pilot Clinical Trial
Brief Title: Biomarker Feedback to Motivate Cessation in Pregnancy
Acronym: MAW Phase 3
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Mayo Clinic (Other)
Collaborators: Alaska Native Tribal Health Consortium (Other); University of California, San Francisco (Other); University of Minnesota (Other)
Responsible Party: Principal Investigator, Christi Patten, PI, Mayo Clinic
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 11-001144-02
Record Dates: First submitted 2015-04-14; First posted 2015-05-01 (Estimated); Last update posted 2017-12-19 (Actual); Status verified 2017-12

CONDITIONS: Nicotine Dependence; Pregnancy
MeSH Terms: conditions — Tobacco Use Disorder

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Control condition (Active Comparator): Control behavioral phone-based smoking cessation intervention
  Interventions: Behavioral: Control condition (phone based smoking cessation counseling)
- Biomarker Feedback Intervention (Experimental): Biomarker feedback plus behavioral phone-based smoking cessation intervention
  Interventions: Behavioral: Biomarker feedback (phone based smoking cessation counseling)

INTERVENTIONS:
Behavioral: Biomarker feedback (phone based smoking cessation counseling) — Feedback on maternal cotinine and likely infant NNAL Phone based behavioral smoking cessation counseling
  Arms: Biomarker Feedback Intervention
Behavioral: Control condition (phone based smoking cessation counseling) — phone-based behavioral smoking cessation counseling
  Arms: Control condition

SUMMARY:
Phase 3 Pilot Clinical Trial.

DETAILED DESCRIPTION:
Developing effective tobacco cessation interventions during pregnancy for American Indian and Alaska Native people is a national priority and will contribute to the U.S. public health objective of reducing tobacco-related cancer health disparities. The proposed project builds on the investigators' successful partnership with the Alaska Native community and previous work with Alaska Native pregnant women. The investigators propose to develop and test a novel biomarker feedback intervention relating cotinine levels in the urine of pregnant women with the woman and infant's likely exposure to the tobacco specific nitrosamine and carcinogen 4-(methylnitrosamino)-1-(3-pyridyl)-1-butanone) (NNK). This 5-year project will be conducted in three phases. In Phase 1 the investigators will utilize a non-randomized, clinical observational trial to examine biomarkers of nicotine and carcinogen exposure (urine cotinine and total NNAL [a metabolite of NNK], respectively) among 150 maternal-infant pairs with assessments conducted during pregnancy and at delivery. In Phase 2, the investigators will obtain qualitative feedback on the findings from Phase 1 through individual interviews conducted with 32 women who use tobacco to develop the biomarker feedback intervention messages. Phase 3 will consist of a formative evaluation of the biomarker feedback intervention with 60 pregnant women using a two-group randomized design to assess the intervention's feasibility and acceptability, and the biochemically confirmed abstinence rate at the end of pregnancy. All phases of the project will be guided by a Community Advisory Committee. Each phase is an important step to advance the investigators' understanding of the potential for biomarker feedback as a strategy to help Alaska Native pregnant women quit tobacco use. The potential reach of the intervention is significant from a public health perspective as over 600 tobacco users deliver each year at the Alaska Native Medical Center in Anchorage where the proposed project will take place. Developing effective interventions for tobacco cessation during pregnancy is important to reduce adverse health consequences for the mother and neonate and future risk of tobacco-caused cancers.

This is the third and final phase of the project.

ELIGIBILITY:
Inclusion Criteria:

* Alaska Native
* 18 years or older
* provide written informed consent
* be currently pregnant and at <24 weeks gestation
* reside in Anchorage and plan to deliver at the ANMC
* current tobacco user defined as any use of Iqmik, commercial ST, and/or cigarettes during the past 7 days.

Exclusion Criteria:

* use of using nicotine replacement therapy or medications for tobacco cessation or participation in a behavioral cessation program within the past 30 days
* another woman from the same household has enrolled.

Ages: 18 Years to 45 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 60 (Actual)
Dates: Start 2015-03; Primary Completion 2017-12 (Actual); Study Completion 2017-12 (Actual)

PRIMARY OUTCOMES:
smoking abstinence in late pregnancy (self-reported abstinence verified with cotinine) | at week 36 gestation or greater up to the time of delivery
  self-reported abstinence verified with cotinine

SECONDARY OUTCOMES:
Self-efficacy (Self-reported confidence scale) | at week 36 gestation or greater up to the time of delivery
  Self-reported confidence scale

CONTACTS AND LOCATIONS:
Overall Officials: Christi A Patten, PhD, Principal Investigator — Mayo Clinic
Locations (1):
- Alaska Native Tribal Health Consortium, Anchorage, Alaska, United States

IPD SHARING:
Plan to Share IPD: No